CLINICAL TRIAL: NCT05634980
Title: The Application of Standardized Dysphagia Diet in Clinical Evaluation of Swallowing Function in Dysphagia Patients
Brief Title: Standardized Dysphagia Diet in Clinical Evaluation of Swallowing Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202105007RINB
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Dysphagia, Swallowing Function, Diet Modification, Dysphagia Diet, Diet Standardization
MeSH Terms: conditions — Deglutition Disorders | interventions — Fees and Charges

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: FEES — Fiberoptic Endoscopic Evaluation of Swallowing (FEES) exam

SUMMARY:
Diet modification has been a vital component in the management of dysphagia. The lingual manipulation of bolus, pharyngeal propulsion, and initiation of swallowing reflex are all affected by the texture of bolus. However, there is a limited literature and consensus regarding how to apply different food consistency in the swallowing function evaluation of dysphagic patients. Recently, International Dysphagia Diet Standardization Initiative (IDDSI) has provided a universal standard of food consistency. The present study aims to evaluate the accuracy of clinical swallowing evaluation using IDDSI standardized food in dysphagic patients, in an attempt to establish protocols of clinical evaluation and diet selection in dysphagic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 years or older with a swallowing disorder on the Functional Oral Intake Scale (FOIS) of 1-6.

Exclusion Criteria:

* Unconscious, unable to communicate via gestures or words and cooperate with commands.
* Acutely infected or requiring respirator use.
* The oropharyngeal structure is abnormal and cannot be examined by endoscopy.
* Presence of tracheostomy tube

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a swallowing disorder
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-08-03 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Penetration aspiration scale (PAS) | Day 1
  Penetration aspiration scale

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan